CLINICAL TRIAL: NCT04335058
Title: Lactoferrin With Iron Versus Iron Alone in Treatment of Anemia In Chronic Liver Disease
Brief Title: Lactoferrin in Treatment of Fe Deficient Anemia In Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/11/2019/1596
Record Dates: First submitted 2020-03-23; First posted 2020-04-06 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Iron Deficiency Anemia; Chronic Liver Failure
MeSH Terms: conditions — Anemia, Iron-Deficiency; End Stage Liver Disease | interventions — Lactoferrin; Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Lactoferrin plus oral iron (Experimental): Treated for 2 months regularly with oral administration of 100 mg Lactoferrin tablet twice a day before meals with oral administration of 100 mg of elemental iron capsules, one capsule twice daily on an empty stomach, at least 1 hour before or 2 hours after meals
  Interventions: Drug: Lactoferrin + Iron Supplement
- Oral iron alone (Active Comparator): Oral administration of 100 mg of elemental iron capsules, one capsule twice daily on an empty stomach, at least 1 hour before or 2 hours after meals
  Interventions: Drug: Iron Supplement

INTERVENTIONS:
Drug: Lactoferrin + Iron Supplement — Lactoferrin 100 mg twice daily +oral iron
  Arms: Group A: Lactoferrin plus oral iron
Drug: Iron Supplement — Oral iron supplement alone
  Arms: Oral iron alone

SUMMARY:
Iron deficiency and altered homeostasis due to inflammation and decreased iron utilization are main factors involved in anemia in liver disease. Lactoferrin is a first line defence protein for protection against microbial infections and subsequent development of systemic disease as seen with systemic inflammatory response syndrome (SIRS) and sepsis. Lactoferrin with iron has been shown to be efficacious with anemia in chronic disease, in pregnancy and in cancer patients with fewer side effects than oral iron alone. High exposure to iron is associated with increased inflammation which is associated with worse cardiovascular outcomes. Lactoferrin can help reduce the total iron dose and hepatic inflammation.

DETAILED DESCRIPTION:
Lactoferrin is a highly conserved, monomeric 80 kDa single polypeptide chain contained in most mammalian exocrine secretions, such as milk, saliva and tears, bronchial, and intestinal secretions. LTF is also found in the secondary granules of neutrophils a glycoprotein present in milk, has been demonstrated to possess a multitude of biological functions. Lactoferrin in Inflammation and Sepsis The antimicrobial activity of LTF is well documented and consists of two mechanisms: one is iron dependent and deals with high affinity of LTF to iron (bacteriostatic), and the other one is due to LTF affinity to lipopolysaccharide (LPS) to function as a direct bactericidal agent for Gram-negative organisms. Small changes, such as single nucleotide polymorphisms, can affect outcomes against pathogenic agents . LTF interacts with cell surface receptors involved in "danger signal" recognition [e.g., toll-like receptor (TLR)4, CD14, and CD22]. At the molecular level, LTF seems to reduce LPS-induced monocyte activation and subsequent production of pro-inflammatory mediators. Lactoferrin in Anemia in Liver Disease The hepatic expression of the hepcidin gene is regulated by signals which reflect body iron status and erythropoietic activity. The regulation of hepcidin by iron status includes a signal from the circulating transferrin via hepatocellular transferrin receptor (TfR2). Like transferrin, lactoferrin will deliver iron to hepatocytes but unlike transferrin, lactoferrin cannot deliver iron to erythroid cells. Lactoferrin does not interact with TfR1 or TfR2.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Either gender
3. Patients with chronic liver disease with iron deficiency anemia with transferrin saturation<20% and Hemoglobin in Non-pregnant women (15 years of age and above) <12g/dl and in men <13g/dl -

Exclusion Criteria:

1. Those who do not consent to participate in the study
2. Inability to obtain informed consent from patient or relatives
3. Severe preexisting cardiopulmonary disease
4. Renal dysfunction (S. Creatinine ≥ 2mg/dL)
5. Pregnancy/Lactation
6. Post liver transplant patients
7. HIV infection
8. Patients who are on psychoactive drugs, like sedatives or antidepressants
9. Patients who are too sick to carry out the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Correction of Anemia | 1 months
  Number of participants achieving Hemoglobin level > 12 g/dl iron deficiency anemia in patients with Chronic Liver Disease of any etiology.
Correction of Anemia | 3 months
  Number of participants achieving Hemoglobin level > 12 g/dl

SECONDARY OUTCOMES:
Reduction in Inflammatory markers | 3 months
  IL-1, Hepcidin, Transferrin saturation measured

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Background] Iwasa M, Kaito M, Ikoma J, Takeo M, Imoto I, Adachi Y, Yamauchi K, Koizumi R, Teraguchi S. Lactoferrin inhibits hepatitis C virus viremia in chronic hepatitis C patients with high viral loads and HCV genotype 1b. Am J Gastroenterol. 2002 Mar;97(3):766-7. doi: 10.1111/j.1572-0241.2002.05573.x. No abstract available. PMID 11922584
- [Background] Actor JK, Hwang SA, Kruzel ML. Lactoferrin as a natural immune modulator. Curr Pharm Des. 2009;15(17):1956-73. doi: 10.2174/138161209788453202. PMID 19519436
- [Background] Elif M, Cooper JA. Upregulation Of Hepcidin Expression By Lactoferrin Administration To Pre-Weanling Mice. Blood, (2013) 122(21), 964.Accessed August 22, 2019.
- [Background] Manzoni P, Rinaldi M, Cattani S, Pugni L, Romeo MG, Messner H, Stolfi I, Decembrino L, Laforgia N, Vagnarelli F, Memo L, Bordignon L, Saia OS, Maule M, Gallo E, Mostert M, Magnani C, Quercia M, Bollani L, Pedicino R, Renzullo L, Betta P, Mosca F, Ferrari F, Magaldi R, Stronati M, Farina D; Italian Task Force for the Study and Prevention of Neonatal Fungal Infections, Italian Society of Neonatology. Bovine lactoferrin supplementation for prevention of late-onset sepsis in very low-birth-weight neonates: a randomized trial. JAMA. 2009 Oct 7;302(13):1421-8. doi: 10.1001/jama.2009.1403. PMID 19809023
- [Background] Hayakawa T, Jin CX, Ko SB, Kitagawa M, Ishiguro H. Lactoferrin in gastrointestinal disease. Intern Med. 2009;48(15):1251-4. doi: 10.2169/internalmedicine.48.2199. Epub 2009 Aug 3. PMID 19652425
- [Background] Lepanto MS, Rosa L, Cutone A, Conte MP, Paesano R, Valenti P. Efficacy of Lactoferrin Oral Administration in the Treatment of Anemia and Anemia of Inflammation in Pregnant and Non-pregnant Women: An Interventional Study. Front Immunol. 2018 Sep 21;9:2123. doi: 10.3389/fimmu.2018.02123. eCollection 2018. PMID 30298070